CLINICAL TRIAL: NCT07001592
Title: A Phase I Dose-Escalation Trial of vvDD-hIL2-2-RG-1 (Vaccina Virus Double Deleted) Administered by Intra-tumoral (IT) Injection for Metastatic Gastrointestinal and Peritoneal Tumors
Brief Title: Intra-tumoral (IT) Injection of vvDD-hIL2-2-RG-1 for Metastatic Gastrointestinal and Peritoneal Tumors
Acronym: RIOT3
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Patrick Wagner, MD, FACS, Director, AHNCI Division of Complex General Surgical Oncology, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIOT3 - vvDD-hIL2-2-RG-1; 2024-087 (Other: AHN Research Institute)
Record Dates: First submitted 2025-05-06; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Gastric Neoplasms; Esophageal Cancer; Liver Cancer; Liver Metastasis; MSS-CRC; MSS; Gastric Adenocarcinoma; Peritoneal Cancer; Peritoneal Carcinoma; Peritoneal Metastases; MSI-H; Gastric Cancer
Keywords: Oncolytic virus; vaccinia; immunotherapy; intra-tumoral; intra-peritoneal
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Vaccinia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- vvDD-hIL-2-RG-1 (Experimental): vvDD-hIL-2-RG-1 administered via intra-tumoral (IT) injection
  Interventions: Biological: vvDD-hIL-2-RG-1

INTERVENTIONS:
Biological: vvDD-hIL-2-RG-1 — A single dose of the investigational agent will be injected intratumorally at one of the following three dose levels.
  Level 1: 3 x 108 p.f.u. Level 2: 1 x 109 p.f.u. Level 3: 3 x 109 p.f.u. p.f.u = Plaque-forming unit(s)
  Dose will be escalated in cohorts of 3, according to a standard 3+3 design.

SUMMARY:
This research study aims to evaluate the safety and determine the optimal dose of a new experimental drug, vvDD-hIL2 (vaccinia virus double-deleted human interleukin 2), in patients with advanced abdominal cancer. The study will involve three dose levels, with three to six patients enrolled at each level.

vvDD-hIL2 is a genetically modified vaccinia virus, derived from the virus previously used for smallpox vaccination. The modification is intended to target and destroy tumors while minimizing harm to healthy tissues by stimulating the body's immune response.

Participants will receive an injection of vvDD-hIL2 directly into their abdominal tumors at AHN West Penn. The study team will monitor for side effects and assess tumor response to the treatment.

Active participation will last up to two months, involving seven clinic visits and approximately four lab visits at AHN West Penn Hospital. Visits will include standard of care procedures as well as study-specific tests and exams. Most visits will last one to two hours, with some extending to two to three hours. The drug administration day will require a twelve-hour visit.

Effectiveness and side effects will be evaluated through blood draws, oral swabs, urinalysis and tissue biopsies. Tissue samples will be used for genomic analysis and stored for potential future research. Data collected may also be used for future research purposes.

Previous human trials of vvDD-hIL2 have reported side effects such as pain, rash or inflammation at the injection site, low-grade fevers, flu-like symptoms, and fatigue. There is a rare risk of rash transmission to close contacts with skin openings, and information on limiting contact and managing rash development will be provided.

DETAILED DESCRIPTION:
This is a Phase I, open-label, single dose, dose-escalation trial in subjects with metastatic gastrointestinal tumors who have failed standard systemic chemotherapy or immunotherapy. Gastrointestinal tumors include esophageal cancer (EC), gastric cancer (GC), colon cancer (CC), rectal cancer (RC), liver cancer (LC), and pancreatic cancer (PC)

The vvDD-IL-2 virus was designed to activate T-cells with a goal to reduce systemic toxicity while optimizing immune clearance of tumors following intraperitoneal delivery. Utilizing a platform of a thymidine kinase (tk) and vaccinia growth factor (vgf) deleted oncolytic Western Reserve (WR) strain vaccinia virus (vvDD), vvDD-IL-2 variants have been designed to deliver membrane bound IL-2 into the tumor microenvironment.

All subjects who have refractory tumors will receive the virus at one of the three dose levels in a single dose sequential dose modified toxicity probability interval (mTPI) design. Eligible subjects will receive one needle injection (per tumor) of vvDD-hIL-2-RG-1. A minimum of 28 days observation period must pass after injection of the first subject in each level without experiencing a dose-limiting toxicity (DLT) before administering/injecting the second patient at that dose level. A new dose level will not be initiated until the completion of the 28-day observation period from the administration of the previous dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age, 18 to < 70 years at the time of consent
2. Histologically confirmed metastases from gastrointestinal tumors with molecular determinants for MSI and KRAS.
3. For microsatellite stable (MSS) tumors, subjects must have failed (or be ineligible for) standard 1st and 2nd line chemotherapy. For microsatellite instability-high (MSI-H) tumors, subjects must also have failed (or be ineligible for) systemic immunotherapy.
4. Karnofsky Performance Status (KPS) of > 70
5. Anticipated survival of at least 12 weeks.
6. Written informed consent in accordance with national, local, and institutional guidelines obtained prior to any study procedures (subject or subject's legally authorized representative (LAR) must have the ability to understand and willingness to sign a written informed consent).
7. Adequate bone marrow function: WBC > 2,000 and <50,000 cells/mm3, ANC > 1,000 cells/mm3, hemoglobin >8 g/dL, and platelet count >100,000 cells/mm3.
8. Adequate renal function: serum creatinine level ≤ 2xULN
9. Adequate liver function: Serum bilirubin < 1.5 x ULN
10. Acceptable coagulation status: INR < ULN +15%. All patients must be able to suspend anticoagulant therapy for study specific biopsies and intra-tumoral injection.
11. Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) must have negative serum or urine pregnancy test.
12. If sexually active, to prevent pregnancy and to prevent the spread of virus, subject must use an acceptable method of contraception as well as barrier contraception from screening through 6 weeks following study treatment with vvDD-hIL-2-RG-1.
13. Subjects must be willing to comply with all study procedures, requirements, adhere to post-treatment care instructions and follow-up examinations.
14. Have measurable disease based on RECIST 1.1 criteria.
15. Have at least one tumor at least 1 cm in diameter amenable to safe intra-tumoral injection.

Exclusion Criteria:

1. Pregnant or nursing an infant.
2. Systemic corticosteroid or other immunosuppressive medication use within 2 weeks of the study treatment.
3. Significant immunodeficiency (e.g. due to underlying illness and/or medication) in subject or household contacts (must be able to avoid household contact with immunodeficient person for 3 weeks).
4. Clinically significant active infection or uncontrolled medical condition (e.g., pulmonary, neurological, cardiovascular, gastrointestinal, genitourinary) considered high risk for investigational new drug treatment, per investigator discretion.
5. Active eczema or psoriasis or other inflammatory skin conditions
6. Unstable cardiac disease which includes but is not limited to any of the following within 6 months prior to study entry: myocardial infarction (MI), unstable angina, congestive heart failure, myocarditis, ventricular arrhythmias diagnosed and requiring medication.

   * New York Heart Association functional class III-IV heart failure on active treatment
   * Pulse oximetry of < 90% in room air at rest
7. Subjects who have received radiation, chemotherapy or other potentially immunosuppressive therapy within 2 weeks prior to study screening and within 4 weeks prior to anticipated vvDD-hIL-2-RG-1 treatment.
8. Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination.
9. Subjects who, in the opinion of the Investigator, have a medical condition that would subject the subject to prohibitive risk by participation in this study, or who may be unable to safely complete the required tumor biopsies.
10. Subjects with household contacts who are children < 5 years old, have active eczema, psoriasis or other inflammatory skin conditions or have a significant immunodeficiency due to underlying illness (e.g. human immunodeficiency virus) and/or medication (e.g. systemic corticosteroids) will be excluded unless alternate living arrangements can be made during the subject's active dosing period and for three weeks following the study medication.
11. Vaccination with a live virus in the previous 60 days prior to Day 0.
12. Inability or unwillingness to give informed consent.
13. Is unable or unwilling to comply with protocol follow-up requirements. -

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety) of vvDD-hIL-2-RG-1 | maximum 28 days
  Measured by frequency and severity of adverse events (AEs) at each dose level as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Maximally-tolerated dose (MTD) of vvDD-hIL-2-RG-1 | maximum 28 days
  Determined by measuring the number of AEs and DLTs at each dose level
Maximum-feasible dose (MFD) of vvDD-hIL-2-RG-1 | maximum 28 days
  Determined by measuring the number of AEs and DLTs at each dose level

SECONDARY OUTCOMES:
Determine the replication rate of vvDD-hIL-2-RG-1 following IT injection | maximum 28 days
  Measured by virus replication in biospecimens (blood, tumor tissue, oral swabs, urine samples and swabs of any skin lesions)
Determine changes in cytokine concentrations and immune cell populations in blood and tissue following vvDD-hIL-2-RG-1 injection using magnetic bead flow cytometry-based assays | maximum 28 days
  Measured by examining concentrations of a panel cytokines and density of immune cell subpopulations in blood and tissue following vvDD-hIL-2-RG-1 injection

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wagner, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- AHN West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No